CLINICAL TRIAL: NCT07025915
Title: A Mass Balance Study of [14C]SSS17 in Healthy Chinese Male Subjects
Brief Title: A Phase 1 Mass Balance Study of [¹⁴C]SSS17 in Healthy Chinese Males
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SSS17-104
Record Dates: First submitted 2025-06-06; First posted 2025-06-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects (HS)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SSS17 (Experimental)
  Interventions: Drug: [14C]SSS17

INTERVENTIONS:
Drug: [14C]SSS17 — single oral dose

SUMMARY:
This study aims to evaluate the absorption, metabolism, and excretion of a single oral dose of [¹⁴C]SSS17 in healthy adult Chinese male subjects, elucidating its overall pharmacokinetic profile in humans to provide essential information for its rational clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male subjects aged 18-45 years .
2. Body weight ≥50 kg .
3. Normal findings on comprehensive health assessment.
4. The subject demonstrates understanding of the trial's objectives, requirements, procedures, and potential adverse reactions; voluntarily participates; commits to complete all trial activities per protocol and comply with study regulations; with the informed consent process conducted in compliance with Good Clinical Practice ."

Exclusion Criteria:

1. Subjects with abnormalities in the nervous system, respiratory system, cardiovascular system, digestive system, hematological and lymphatic systems, endocrine system, or musculoskeletal system that are deemed clinically significant by the investigator.
2. History of organic heart disease
3. History of hypersensitivity or allergy to active ingredients.
4. Average daily smoking >5 cigarettes within 3 months prior to screening or inability to abstain during the trial.
5. Average weekly alcohol intake >14 units within 3 months prior to screening or positive alcohol breath test.
6. History of drug abuse or illicit drug use, or positive urine drug screen.
7. Participation in any other investigational drug trial within 3 months prior to screening.
8. Use of any prescription/non-prescription medication within 2 weeks prior to investigational product administration.
9. History of needle/phobia or inability to tolerate venipuncture.
10. Hemorrhoids/active perianal bleeding, chronic constipation/diarrhea or positive fecal occult blood test at screening.
11. Occupational radiation exposure;
12. Pregnancy plans during or within 1 year post-trial, or refusal to use strict contraception by subject/partner during and within 1 year post-trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Cumulative excretion rate of radioactivity in excreta (urine, feces) and total radioactivity (urine and feces) | up to Day 22
Cmax | up to day22
Tmax | up to Day22

SECONDARY OUTCOMES:
AEs | up to day 22

IPD SHARING:
Plan to Share IPD: Undecided